CLINICAL TRIAL: NCT03510624
Title: Investigation of the Acute Effect of Rebaudioside A on the Glucose Excursion During an Oral Glucose Tolerance Test in 30 Patients With Type 2 Diabetes Mellitus (AREBAG)
Brief Title: Acute Effect of Rebaudioside A on Glucose Excursion During an Oral Glucose Tolerance Test in Type 2 Diabetes Mellitus
Acronym: AREBAG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: s61580
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rebaudioside A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First rebaudioside A and then placebo (Experimental)
  Interventions: Drug: Rebaudioside A; Drug: Placebo
- First placebo and then rebaudioside A (Experimental)
  Interventions: Drug: Rebaudioside A; Drug: Placebo

INTERVENTIONS:
Drug: Rebaudioside A — Rebaudioside A 3g
Drug: Placebo — Empty capsules

SUMMARY:
Investigate the acute effect of the steviol glycoside, rebaudioside A, on the glucose excursion during an oral glucose tolerance test in 30 patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Eligible individuals with type 2 diabetes mellitus will be invited for four study visits. During the first and third study visit, rebaudioside A or the placebo will be administered. During the second and fourth study visit, an oral glucose tolerance test (OGTT) will be executed to measure the response of administration of rebaudioside A versus placebo on the glucose homeostasis. The area under the curve blood glucose values during the first two hours of the OGTT will be compared for both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent
* Understand procedures
* Type 2 diabetes mellitus
* Body Mass Index (BMI): 25 - 40 kg/m2
* HbA1c: 6.5-8%
* Judged to be in good health

Exclusion Criteria:

* Subject is unable to

  * Refrain from stevia leaves, stevia extracts or steviol glycoside-containing products from 5 days prior to administration of rebaudioside A or placebo until discharge from the unit after the OGTT on the consecutive day.
  * Refrain from quinine-containing products from 72h prior to administration of rebaudioside A or placebo until discharge from the unit after the OGTT on the consecutive day.
  * Maintain their habitual diets and physical activity patterns and refrain from engaging in strenuous physical activities from 72h prior to administration of rebaudioside A or placebo until discharge from the unit after the OGTT on the consecutive day.
  * Refrain from grapefruit products from 14 days before study visit 1 until discharge from the unit after the OGTT on study visit 4.
  * Refrain from alcohol from 24h prior to administration of rebaudioside A or placebo until discharge from the unit after the OGTT on the consecutive day.
  * Refrain from caffeine containing products from 12h prior to administration of rebaudioside A or placebo until discharge from the unit after the OGTT on the consecutive day.
  * Fast at least 5 hours prior to the administration of rebaudioside A or placebo on study days 1 and 3.
  * Fast at least 10 hours prior to the study days 2 and 4.
* Women of childbearing potential (last menstruation less than 1 year prior to screening) who are pregnant, lactating or planning to become pregnant during the study.
* Individuals with other forms of diabetes
* Current or previous treatment with any diabetes drug within 3 months prior to screening, except for metformin.
* Symptomatic hyperglycemia requiring immediate therapy during screening, in the judgement of the principal investigator.
* Evidence of significant diabetic complications.
* History of pancreas or beta-cell transplantation.
* Presence or history of clinically relevant medical, surgical or psychiatric conditions likely to affect the subject's safety in this trial or that could confound the study assessments or endpoints.
* Clinically relevant abnormal physical findings.
* Clinically significant abnormalities of vital signs:

  * Seated systolic blood pressure outside 90-160 mmHg
  * Diastolic blood pressure outside 40-100 mmHg
  * Heart rate <50 bpm
  * Corrected QT (QTC) using Fridericia's formulae >450 msec (for men) or >470 msec (for women) measured with a 12-lead electrocardiogram.
  * Clinically significant abnormal laboratory values.
  * Moderate or severe renal dysfunction defined as a calculated glomerular filtration rate (GFR) <30 ml/min.
* Currently active or history of alcohol abuse.
* Currently active or history of drug addiction or currently a regular user of drugs including "recreational use" of any illicit drug.
* Smoking cigarettes or using nicotine-containing products, during the last 6 months prior to screening, as nicotine inhibits the Transient Receptor Potential 5 (TRPM5) channel.
* Individuals for whom a major surgery is planned to occur between screening and the end of the trial.
* Previous or current use of concomitant medication, which would confound the study conduct or implicate a risk for safety of the participant, as judged by the investigator(s).
* History of relevant drug or food allergies or a history of severe anaphylactic reaction.
* History of hypersensitivity to the study drug or any of the excipients or to medicinal products with similar chemical structures.
* Individuals with hepatitis B and/or hepatitis C virus.
* Individuals with Human Immunodeficiency Virus (HIV).
* Participation in another clinical trial involving an investigational product within the 3 months preceding screening or 5-halflives of the drug studied, whichever is longer, prior to study supplement administration. Or, participation in any other type of medical research within 3 months preceding screening judged not to be scientifically or medically compatible with this study.
* Individuals who have donated or lost more than 500 ml blood or plasma within 3 months prior to screening.
* Individuals unable to swallow orally administered medication.
* Individuals in which catheter placement is impossible (amputation, no visible veins, …)
* Individuals that cannot speak or understand the Dutch language.
* In the opinion of the principal investigator any other factor that could interfere with the subject's ability to provide informed consent or to complete the study with strict compliance to the study protocol, or that could hold safety concerns for the subject or could impact the outcome of the study results.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) blood glucose concentrations during an OGTT | 0 to 2 hours after glucose challenge
  Area under the curve blood glucose concentrations during an OGTT

SECONDARY OUTCOMES:
AUC glucose/insulin/glucagon | -30 to 0 min of OGTT
  AUC glucose/insulin/glucagon
AUC glucose/insulin/glucagon | 0 to 30 min of OGTT
  AUC glucose/insulin/glucagon
AUC glucose/insulin/glucagon | 0 to 4 hours of OGTT
  AUC glucose/insulin/glucagon
Maximal blood glucose | -30 min to 4 hours of OGTT
  Maximal blood glucose
Maximal blood glucose excursion | -30 min to 4 hours of OGTT
  Maximal blood glucose excursion
Maximal serum insulin | -30 min to 4 hours of OGTT
  Maximal serum insulin
Maximal serum glucagon | -30 min to 4 hours of OGTT
  Maximal serum glucagon
Concentration(t) (C(t))rebaudioside A, steviol and steviol glucuronide | -30 min to 4 hours of OGTT
  Concentration of rebaudioside A, steviol and steviol glucuronide on different time points

CONTACTS AND LOCATIONS:
Overall Officials: Bart Van der Schueren, Principal Investigator — UZ Leuven
Locations (1):
- Centrum Clinical Pharmacology, Leuven, Flanders, Belgium

REFERENCES:
- [Derived] Simoens C, Philippaert K, Wuyts C, Goscinny S, Van Hoeck E, Van Loco J, Billen J, de Hoon J, Ampe E, Vangoitsenhoven R, Mertens A, Vennekens R, Van der Schueren B. Pharmacokinetics of Oral Rebaudioside A in Patients with Type 2 Diabetes Mellitus and Its Effects on Glucose Homeostasis: A Placebo-Controlled Crossover Trial. Eur J Drug Metab Pharmacokinet. 2022 Nov;47(6):827-839. doi: 10.1007/s13318-022-00792-7. Epub 2022 Sep 3. PMID 36057030